CLINICAL TRIAL: NCT04671667
Title: A Phase II Randomized Trial of Adjuvant Therapy With Pembrolizumab After Resection of Recurrent/Second Primary Head and Neck Squamous Cell Carcinoma With High Risk Features
Brief Title: Testing What Happens When an Immunotherapy Drug (Pembrolizumab) is Given by Itself Compared to the Usual Treatment of Chemotherapy With Radiation After Surgery for Recurrent Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-13174; NCI-2020-13174 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA3191 (Other: ECOG-ACRIN Cancer Research Group); EA3191 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2020-12-16; First posted 2020-12-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Oral Cavity Squamous Cell Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; pembrolizumab; Proton Therapy; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm B (cisplatin, carboplatin, IMRT, PBRT) (Active Comparator): Patients receive cisplatin or carboplatin IV on day 1. Treatment repeats every 7 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo IMRT or PBRT QD for a total of 30 fractions in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI throughout the trial.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Radiation: Proton Beam Radiation Therapy
- Arm C (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 6 weeks for 9 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI throughout the trial.
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm B (cisplatin, carboplatin, IMRT, PBRT)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm B (cisplatin, carboplatin, IMRT, PBRT)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
  Arms: Arm B (cisplatin, carboplatin, IMRT, PBRT)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
  Arms: Arm C (pembrolizumab)
Radiation: Proton Beam Radiation Therapy — Undergo PBRT
  Other Names: External beam radiation therapy protons (procedure); External Beam Radiotherapy (protons); PBRT; Proton; Proton EBRT; Proton External Beam Radiotherapy; Proton Radiation Therapy; PROTON Therapy; Radiation, Proton Beam
  Arms: Arm B (cisplatin, carboplatin, IMRT, PBRT)

SUMMARY:
This phase II trial studies the effect of pembrolizumab alone compared to the usual approach (chemotherapy [cisplatin and carboplatin] plus radiation therapy) after surgery in treating patients with head and neck squamous cell carcinoma that has come back (recurrent) or patients with a second head and neck cancer that is not from metastasis (primary). Radiation therapy uses high energy radiation or protons to kill tumor cells and shrink tumors. Cisplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of cancer cells. Carboplatin is also in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of cancer cells. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer and may interfere with the ability of tumor cells to grow and spread. Giving pembrolizumab alone after surgery may work better than the usual approach in shrinking recurrent or primary head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate overall survival (OS) of adjuvant pembrolizumab for 12 months compared to adjuvant reirradiation plus concurrent platinum chemotherapy in high risk head and neck squamous cell carcinoma (HNSCC) patients.

SECONDARY OBJECTIVES:

I. To evaluate the following endpoints in both arms: disease free survival (DFS), locoregional control, rates of distant metastasis, toxicity.

II. To evaluate whether high PD-L1 expression (defined as Combined Positive Score [CPS] >= 20) is predictive of increased efficacy in the experimental group compared to control.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM B: Patients receive cisplatin or carboplatin intravenously (IV) on day 1. Treatment repeats every 7 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo intensity-modulated radiation therapy (IMRT) or proton beam radiation therapy (PBRT) once daily (QD) for a total of 30 fractions in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 6 weeks for 9 cycles in the absence of disease progression or unacceptable toxicity.

Patients in all arms undergo computed tomography (CT) or magnetic resonance imaging (MRI) throughout the trial.

After completion of study treatment, patients are followed up at 30 days, and then every 6 months for up to 5 years from the date of registration.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be between 18 and 79 years of age
* Patient must have locoregionally recurrent or second primary HNSCC (oral cavity, oropharynx, larynx, hypopharynx) in a previously radiated field
* Patient must have undergone surgery with gross total resection and must be randomized within 8 weeks of surgery
* Patients must have high risk disease defined as:

  * Positive margins and/or extra nodal extension (ENE)

    * Positive margins are defined as malignancy at or within 1 mm of the margin. High grade dysplasia (i.e. carcinoma in situ) at the margin is also considered positive
    * ENE may be either gross or microscopic
* Patient must have a PD-L1 Combined Positive Score (CPS) >= 1 in a Clinical Laboratory Improvement Act (CLIA) certified laboratory. Testing can be done locally as long as it is done in a CLIA certified laboratory. This testing must be on the tumor specimen from the resection of the patient's recurrent or second primary HNSCC
* Patient must have had prior radiation to the area of recurrent or second primary tumor. This is defined as > 50% of the presurgical tumor volume having previously received a dose of > 45 Gy as determined by the treating radiation oncologist
* Patient must have completed prior radiation a minimum of 6 months prior to randomization
* Patient must not have any evidence of distant disease based on baseline imaging done within 28 days prior to randomization
* Patient must not have received anti-PD-1/PD-L1 therapy for recurrent disease. If the patient received anti-PD-1/PD-L1 therapy as part of initial upfront curative intent treatment (either as part of definitive non-surgical therapy or in the adjuvant setting) in the past, the last dosage of anti-PD-1/PD-L1 therapy must have been given greater than one year prior to randomization
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used. All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy. A urine or serum pregnancy test must be repeated within 72 hours prior to receiving the first dose of pembrolizumab or chemotherapy if the test done for eligibility/randomization is done outside of this 72 hour window. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. A patient of childbearing potential is someone, regardless of whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patient must not expect to conceive or father children by using by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse while on study treatment, and continue for 120 days after the last dose of study treatment
* Absolute neutrophil count (ANC) >= 1,500/mcL (obtained =< 28 days prior to protocol randomization)
* Platelets >= 100,000/mcL (obtained =< 28 days prior to protocol randomization)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (obtained =< 28 days prior to protocol randomization)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3.0 x institutional ULN (obtained =< 28 days prior to protocol randomization)
* Creatinine clearance > 30 ml/min using the Cockcroft-Gault formula (obtained =< 28 days prior to protocol randomization)
* Patient must not have a current active infection that requires systemic treatment at time of randomization
* Patient must not have a history of non-infectious pneumonitis requiring steroids within 3 years prior to randomization
* Patient must not have a history of solid organ transplant or stem cell transplant
* Patient must not be on immunosuppressive medication within 7 days prior to randomization, EXCEPT for the following: a) intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b) systemic corticosteroids at physiologic doses =< 10 mg/day of prednisone or equivalent; c) steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional classification. Patients with New York Heart Association class III or IV heart failure are not eligible
* Patient must not have received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist [registered trademark]) are live attenuated vaccines and are not allowed
* Patient must not have severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients
* Patient must not have an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
* Patient must not have a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial as long as they have not been HIV-infected with a history of Kaposi sarcoma and/or multicentric Castleman disease
* Patient must not have a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV ribonucleic acid [RNA] [qualitative] is detected) infection

  * NOTE: No testing for hepatitis B and hepatitis C is required unless mandated by a local health authority

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization to date of death from any cause, measured at 2 years
  Kaplan-Meier estimates will be used to estimate the OS distributions. A log-rank test with one-sided 10% type I error will be used for the comparison.
Incidence of adverse events | Up to 5 years from date of registration
  Assessed using Common Terminology Criteria for Adverse Events. An 80% confidence interval around the hazard ratio of the two experimental arms will be calculated. Toxicity will be compared between the two treatment arms. Toxicity will be examined by arm and compared using the Fisher's exact test.

SECONDARY OUTCOMES:
Disease free survival | From the date of randomization to the date of recurrence, second primary tumor from the head and neck region, or death, assessed up to 5 years from date of registration
PD-L1 expression | Up to 5 years from date of registration
  Defined as Combined Positive Score >= 20 as a predictive marker of efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Dan P Zandberg, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (170):
- United States (170):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente-Ontario, Ontario, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - California Protons Cancer Therapy Center, San Diego, California
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Reid Health, Richmond, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - UPMC Altoona, Altoona, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Avera Cancer Institute at Yankton, Yankton, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm